CLINICAL TRIAL: NCT07372248
Title: Comparison of the Effects of Different Surgical Techniques on the Degree of Thermal Artifact in Patients Undergoing Conization: A Clinical Study
Brief Title: Thermal Artifact in Patients Undergoing Conization: A Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106751
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Cervix Neoplasm; Cervix, Dysplasia
Keywords: conization
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Conization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pure Cut (Active Comparator): Conization with Electrosurgery: Power Setting 50 watts pure cut
  Interventions: Procedure: Conization with Electrosurgery diffferent power settings
- Blend (Active Comparator): Conization with Electrosurgery:Power Setting 50 watts blend
  Interventions: Procedure: Conization with Electrosurgery diffferent power settings
- Hybrid (Experimental): Conization with Electrosurgery and Knife: Power Setting 50 watts pure cut and knife
  Interventions: Procedure: Conization with Electrosurgery diffferent power settings

INTERVENTIONS:
Procedure: Conization with Electrosurgery diffferent power settings — 50 watts pure cut,50 watts blend mode

SUMMARY:
Cervical transformation zone excision is commonly used in the diagnosis and treatment of cervical intraepithelial neoplasia. Thermal artifacts can negatively affect histopathological evaluation. This study compares three different modifications of conization performed using electrosurgery in terms of the degree of thermal artifacts.

DETAILED DESCRIPTION:
Conization procedures performed using electrosurgical techniques, such as LEEP, NETZ, and SWETZ, are well described in the literature. Compared with cold knife conization, these methods offer several advantages, including the ability to be performed under local anesthesia, shorter procedure time, and lower cost. However, electrosurgical techniques may compromise histopathological evaluation of surgical specimens due to the presence of thermal artifacts, which can obscure tissue architecture and surgical margins.

In our clinic, conization procedures are routinely performed using a hybrid technique that combines electrosurgery with cold knife conization. This study aims to compare three different modifications of this hybrid technique applied in our institution with respect to the degree of thermal artifact formation and the quality of surgical margin evaluation.

ELIGIBILITY:
Inclusion Criteria:Women aged ≥18 years

Indication for LLETZ based on abnormal cervical cytology and/or biopsy

Ability to provide written informed consent -

Exclusion Criteria: Previous cervical excisional procedure

Pregnancy

Active cervical infection

History of cervical cancer

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Thermal Artefact | Within 7 days following the surgical procedure
  Thermal artifact will be assessed by blinded gynecologic pathologists using a structured histopathological evaluation based on epithelial distortion, coagulative necrosis, and interference with margin interpretation. Thermal artifact severity will be graded as none, mild, moderate, or severe.

SECONDARY OUTCOMES:
TZ evaluation | postoperative 4th month
  Transformation zone visibility will be evaluated during postoperative colposcopic examination and categorized as fully visible, partially visible, or not visible.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Bas, Principal Investigator — Universty of Health Science

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prendiville W, Cullimore J, Norman S. Large loop excision of the transformation zone (LLETZ). A new method of management for women with cervical intraepithelial neoplasia. Br J Obstet Gynaecol. 1989 Sep;96(9):1054-60. doi: 10.1111/j.1471-0528.1989.tb03380.x. PMID 2804007
- [Background] Watanabe Y, Fuchshuber P, Homma T, Bilgic E, Madani A, Hiki N, Cammack I, Noji T, Kurashima Y, Shichinohe T, Hirano S. An Unmodulated Very-Low-Voltage Electrosurgical Technology Creates Predictable and Ultimate Tissue Coagulation: From Experimental Data to Clinical Use. Surg Innov. 2020 Oct;27(5):492-498. doi: 10.1177/1553350620904610. Epub 2020 Mar 18. PMID 32186463
- [Background] Nagar HA, Dobbs SP, McClelland HR, Price JH, McClean G, McCluggage WG. The large loop excision of the transformation zone cut or blend thermal artefact study: a randomized controlled trial. Int J Gynecol Cancer. 2004 Nov-Dec;14(6):1108-11. doi: 10.1111/j.1048-891X.2004.14608.x. PMID 15571616